CLINICAL TRIAL: NCT05053607
Title: Clinical and Patient Reported Outcomes for Individuals with Relapsed/Refractory Multiple Myeloma Treated with Isatuximab: Real-World Insights from Patient Reported, Wearable, and Qualitative Data in the Context of Digital Health Coaching
Brief Title: Real World Insights During Treatment for Relapsed/Refractory Multiple Myeloma with Isatuximab
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pack Health (Industry)
Collaborators: M.D. Anderson Cancer Center (Other); Sanofi (Industry); University of Washington (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021-0309
Record Dates: First submitted 2021-09-07; First posted 2021-09-22 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Multiple Myeloma; Refractory Multiple Myeloma
Keywords: isatuximab; wearable electronic devices; qualitative research; patient reported outcome measures
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: A single cohort of 50 individuals with relapsed/refractory multiple myeloma will be enrolled in the study, all of which will be enrolled in a digital health coaching program and receive a Fitbit device for activity tracking. Individuals from both study sites will be enrolled to this single cohort.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 1. Single Arm Cohort Receiving Digital Health Coaching (Other): All study participants will be enrolled in a 3-month digital health coaching program. They will also receive a Fitbit device to be worn daily for the capture of physical activity data.
  Participants have the option to participate in a one time interview about their treatment experience.
  Interventions: Behavioral: Digital Health Coaching Program; Device: Fitbit

INTERVENTIONS:
Behavioral: Digital Health Coaching Program — consisting of weekly calls and delivery of evidence-based content across health and wellness domains (e.g. nutrition, exercise, physical, emotional and financial health) up to 4 times weekly via text, email or mobile application.
Device: Fitbit — A wrist-worn activity tracker allowing for the capture of physical activity, including but not limited to step-count and minutes of activity, to be captured daily.

SUMMARY:
This descriptive study aims to evaluate the experience of adults with relapsed or refractory multiple myeloma receiving standard of care isatuximab-irfc through collection of quantitative, qualitative and wearable data. Fifty adults with relapsed or refractory multiple myeloma receiving standard of care isatuximab-irfc will be enrolled across 2 sites, The University of California San Francisco and The University of Texas MD Anderson Cancer Center. Consented participants will be enrolled in a 3-month digital health coaching program through which electronic patient reported outcomes and wearable activity data will be collected. Outcomes include treatment experience, quality of life, financial toxicity, treatment adherence, symptom burden and health self-efficacy. These will be captured by patient reported outcome measures including the Patient's Qualitative Assessment of Treatment- Real World (PQAT-RW), Patient Global Impression of Change/Severity (PGIC/S), European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-C30), Quality of Life Questionnaire Multiple Myeloma (QLQ-MY20), and the European QoL-5 Dimensions (EQ5D), Cancer Behavior Inventory-Brief Form (CBI-B), Center for Adherence Support Evaluation (CASE) Medication Adherence Index, Comprehensive Score for Financial Toxicity (COST) Instrument.

Clinical data, including treatment history, healthcare utilization, and co-morbidities, as well as demographic data will be collected via the electronic health record from each clinical site. This data will be complemented by qualitative data from a selected cohort of study participants with a focus on treatment experience ranging from infusion burden, toxicity management, to overall quality of life. Evaluation of this data in combination will be used to better understand the treatment experience of individuals on standard of care isatuximab-irfc specifically, and with relapsed or refractory multiple myeloma generally, contributing to an existing gap in the literature regarding patient reported outcomes from diverse data sources. Outcomes will be analyzed with attention to the relationship between social determinants of health, including race, ethnicity, and geographic location, and treatment experience as reflected in both the qualitative and quantitative data.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Diagnosis of relapsed/refractory multiple myeloma corresponding to the Food and Drug Administration (FDA) package insert for isatuximab-irfc (Sarclisa®).
* Confirmed or planned treatment with intravenous isatuximab-irfc for relapsed/refractory multiple myeloma as standard-of-care therapy. Concurrent therapy with other agents (e.g., pomalidomide) is allowed.
* Access to and willingness to use a smartphone or other device through which they can send and receive text messages, emails and/or access a mobile application.
* Willingness to wear and have data collected by a Fitbit
* Ability to engage in physical activity as evidenced by an Eastern Cooperative Oncology Group (ECOG) performance status score of less than or equal to 2

Exclusion Criteria:

* Individuals who are terminally ill, defined as individuals identified by their physician as likely having 6 months or less to live, or those individuals transitioned to comfort measures only (meaning only supportive care measures without curative focused treatment)
* Individuals for whom there is documentation of inability to provide consent in the medical record.
* Individuals receiving isatuximab-irfc subcutaneously

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-06-17 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Patient's Qualitative Assessment of Treatment Real World version (PQAT-RW) | Change in baseline perception of treatment experience at 3 months
  A 6-item survey assessing experience of a drug during clinical trial. The instrument consists of 3-free text and 3 scaled responses assessing the perceived benefits and disadvantages of received treatment and willingness to continue on drug after the study.
Qualitative Interview | Within the last month of study participation
  A one time interview will be conducted to learn more about the experience of individuals related to their diagnosis, treatment, symptoms, side effects and overall care experience.

SECONDARY OUTCOMES:
Change in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-C30) | Change in baseline perception of treatment experience at 3 months
  A 30-item measure of quality of life across 5 domains, including physical, emotional, social, role and cognitive), 8 symptoms, and items assessing global health and financial toxicity. Recall over the past week is scored primarily on a 4-point scale ranging from "not at all" to "very much". The instrument may be administered either on paper or electronically.
Change in Quality of Life Questionnaire Multiple Myeloma (QLQ-MY20) | Change in baseline perception of treatment experience at 3 months
  A 20-item measure of quality of life among individuals with multiple myeloma. It assesses a series of symptoms on a 4-point Likert scale ranging from 1 (Not at All) to 4 (Very Much).
Change in European QoL-5 Dimensions (EQ5D) | Change in baseline perception of treatment experience at 3 months
  A measure of quality of life across 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
Change in Cancer Behavior Inventory-Brief Form (CBI-B) | Change in baseline perception of treatment experience at 3 months
  This 12-item instrument measures self-efficacy in coping with cancer across 7 domains. These include: Seeking and Understanding Medical Information, Emotion Regulation, Coping with Treatment Related Side Effects, Accepting Cancer/ Maintaining a Positive Attitude, Seeking Social Support, and Using Spiritual Coping. The instrument utilizes a 9-point response scale ranging from 1 "Not at all confident" to 9 "Confident".
Change in Patient Global Impression of Severity (PGIS) Scale | Change in baseline perception of treatment experience at 3 months
  A 1-item measure of severity of relapsed/refractory multiple myeloma symptoms since the last visit, which is scored a on a 5-response scale ranging from "none" to "very severe".
Change in Patient Global Impression of Change (PGIC) Scale | Change in baseline perception of treatment experience at 3 months
  A 1-item measure of patient perception of change in relapsed/refractory multiple myeloma symptoms since starting a study. Responses are scored on a 7-point scale, ranging from "very much worse" to "very much better".
Change in Center for Adherence Support Evaluation (CASE) Medication Adherence Index | Change in baseline perception of treatment experience at 3 months
  The Center for Adherence Support Evaluation (CASE) is a three-item questionnaire used to measure antiretroviral therapy adherence. This questionnaire was developed through the Special Projects of National Significance (SPNS) initiative called Assessing Existing Efforts to Increase Adherence to Medication. Patients take less than 5 minutes to answer the three unique questions, asking about their difficulty taking medications on time, average days per week with one dose missed, and the last time they missed a dose.
Change in Comprehensive Score for Financial Toxicity (COST) Instrument | Change in baseline perception of treatment experience at 3 months
  The Comprehensive Score for Financial Toxicity (COST) is an 11-item instrument used to measure the financial toxicity of cancer treatment, which has been demonstrated to be highly correlated with HRQoL (de Souza et al., 2017). This instrument was validated among individuals with advanced cancer and demonstrated high internal consistency (Cronbach's α >.90) and highly correlated to HRQol (p=.05). The instrument consists of 11 items, utilizing a five-point ordinal scale ranging from (0- Not at all) to (4- Very much).

OTHER OUTCOMES:
Physical Activity | From date of enrollment up to 3 months
  Physical activity, including step count and minutes of physical activity will be collected via Fitbits provided to study participants
Health Care Utilization | From date of enrollment up to 3 months
  ER visits and unplanned hospitalizations
Digital Engagement | From date of enrollment up to 3 months
  Frequency, types and duration of engagement with the digital health coaching platform

CONTACTS AND LOCATIONS:
Overall Officials: Melody R Becnel, MD, Principal Investigator — M.D. Anderson Cancer Center; Rahul Banerjee, MD, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Basch E, Deal AM, Dueck AC, Scher HI, Kris MG, Hudis C, Schrag D. Overall Survival Results of a Trial Assessing Patient-Reported Outcomes for Symptom Monitoring During Routine Cancer Treatment. JAMA. 2017 Jul 11;318(2):197-198. doi: 10.1001/jama.2017.7156. PMID 28586821
- [Background] Cocks K, Cohen D, Wisloff F, Sezer O, Lee S, Hippe E, Gimsing P, Turesson I, Hajek R, Smith A, Graham L, Phillips A, Stead M, Velikova G, Brown J; EORTC Quality of Life Group. An international field study of the reliability and validity of a disease-specific questionnaire module (the QLQ-MY20) in assessing the quality of life of patients with multiple myeloma. Eur J Cancer. 2007 Jul;43(11):1670-8. doi: 10.1016/j.ejca.2007.04.022. Epub 2007 Jun 15. PMID 17574838
- [Background] de Souza JA, Yap BJ, Wroblewski K, Blinder V, Araujo FS, Hlubocky FJ, Nicholas LH, O'Connor JM, Brockstein B, Ratain MJ, Daugherty CK, Cella D. Measuring financial toxicity as a clinically relevant patient-reported outcome: The validation of the COmprehensive Score for financial Toxicity (COST). Cancer. 2017 Feb 1;123(3):476-484. doi: 10.1002/cncr.30369. Epub 2016 Oct 7. PMID 27716900
- [Background] Girault A, Ferrua M, Lalloue B, Sicotte C, Fourcade A, Yatim F, Hebert G, Di Palma M, Minvielle E. Internet-based technologies to improve cancer care coordination: current use and attitudes among cancer patients. Eur J Cancer. 2015 Mar;51(4):551-557. doi: 10.1016/j.ejca.2014.12.001. Epub 2015 Feb 4. PMID 25661828
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Heitzmann CA, Merluzzi TV, Jean-Pierre P, Roscoe JA, Kirsh KL, Passik SD. Assessing self-efficacy for coping with cancer: development and psychometric analysis of the brief version of the Cancer Behavior Inventory (CBI-B). Psychooncology. 2011 Mar;20(3):302-12. doi: 10.1002/pon.1735. PMID 20878830
- [Background] Kent EE, Ambs A, Mitchell SA, Clauser SB, Smith AW, Hays RD. Health-related quality of life in older adult survivors of selected cancers: data from the SEER-MHOS linkage. Cancer. 2015 Mar 1;121(5):758-65. doi: 10.1002/cncr.29119. Epub 2014 Nov 4. PMID 25369293
- [Background] Madduri D, Dhodapkar MV, Lonial S, Jagannath S, Cho HJ. SOHO State of the Art Updates and Next Questions: T-Cell-Directed Immune Therapies for Multiple Myeloma: Chimeric Antigen Receptor-Modified T Cells and Bispecific T-Cell-Engaging Agents. Clin Lymphoma Myeloma Leuk. 2019 Sep;19(9):537-544. doi: 10.1016/j.clml.2019.08.002. Epub 2019 Aug 7. PMID 31427259
- [Background] Madore S, Kilbourn K, Valverde P, Borrayo E, Raich P. Feasibility of a psychosocial and patient navigation intervention to improve access to treatment among underserved breast cancer patients. Support Care Cancer. 2014 Aug;22(8):2085-93. doi: 10.1007/s00520-014-2176-5. Epub 2014 Mar 18. PMID 24639035
- [Background] Mannheimer SB, Mukherjee R, Hirschhorn LR, Dougherty J, Celano SA, Ciccarone D, Graham KK, Mantell JE, Mundy LM, Eldred L, Botsko M, Finkelstein R. The CASE adherence index: A novel method for measuring adherence to antiretroviral therapy. AIDS Care. 2006 Oct;18(7):853-61. doi: 10.1080/09540120500465160. PMID 16971298
- [Background] Moreno L, Perez C, Zabaleta A, Manrique I, Alignani D, Ajona D, Blanco L, Lasa M, Maiso P, Rodriguez I, Garate S, Jelinek T, Segura V, Moreno C, Merino J, Rodriguez-Otero P, Panizo C, Prosper F, San-Miguel JF, Paiva B. The Mechanism of Action of the Anti-CD38 Monoclonal Antibody Isatuximab in Multiple Myeloma. Clin Cancer Res. 2019 May 15;25(10):3176-3187. doi: 10.1158/1078-0432.CCR-18-1597. Epub 2019 Jan 28. PMID 30692097
- [Background] Saunders B, Sim J, Kingstone T, Baker S, Waterfield J, Bartlam B, Burroughs H, Jinks C. Saturation in qualitative research: exploring its conceptualization and operationalization. Qual Quant. 2018;52(4):1893-1907. doi: 10.1007/s11135-017-0574-8. Epub 2017 Sep 14. PMID 29937585
- [Background] Thorne S, Kirkham SR, MacDonald-Emes J. Interpretive description: a noncategorical qualitative alternative for developing nursing knowledge. Res Nurs Health. 1997 Apr;20(2):169-77. doi: 10.1002/(sici)1098-240x(199704)20:23.0.co;2-i. PMID 9100747
- [Background] Osoba D, Aaronson N, Zee B, Sprangers M, te Velde A. Modification of the EORTC QLQ-C30 (version 2.0) based on content validity and reliability testing in large samples of patients with cancer. The Study Group on Quality of Life of the EORTC and the Symptom Control and Quality of Life Committees of the NCI of Canada Clinical Trials Group. Qual Life Res. 1997 Mar;6(2):103-8. doi: 10.1023/a:1026429831234. PMID 9161109
- [Background] Pearman TP, Beaumont JL, Mroczek D, O'Connor M, Cella D. Validity and usefulness of a single-item measure of patient-reported bother from side effects of cancer therapy. Cancer. 2018 Mar 1;124(5):991-997. doi: 10.1002/cncr.31133. Epub 2017 Nov 13. PMID 29131323
- [Background] Proskorovsky I, Lewis P, Williams CD, Jordan K, Kyriakou C, Ishak J, Davies FE. Mapping EORTC QLQ-C30 and QLQ-MY20 to EQ-5D in patients with multiple myeloma. Health Qual Life Outcomes. 2014 Mar 11;12:35. doi: 10.1186/1477-7525-12-35. PMID 24618388
- [Background] Ventura F, Ohlen J, Koinberg I. An integrative review of supportive e-health programs in cancer care. Eur J Oncol Nurs. 2013 Aug;17(4):498-507. doi: 10.1016/j.ejon.2012.10.007. Epub 2012 Nov 15. PMID 23158437
- [Background] Zaleta AK, Miller MF, Olson JS, Yuen EYN, LeBlanc TW, Cole CE, McManus S, Buzaglo JS. Symptom Burden, Perceived Control, and Quality of Life Among Patients Living With Multiple Myeloma. J Natl Compr Canc Netw. 2020 Aug;18(8):1087-1095. doi: 10.6004/jnccn.2020.7561. PMID 32755984
- [Background] Zhang T, Wang S, Lin T, Xie J, Zhao L, Liang Z, Li Y, Jiang J. Systematic review and meta-analysis of the efficacy and safety of novel monoclonal antibodies for treatment of relapsed/refractory multiple myeloma. Oncotarget. 2017 May 16;8(20):34001-34017. doi: 10.18632/oncotarget.16987. PMID 28454113